CLINICAL TRIAL: NCT00401245
Title: The Effect of Dose Titration and Dose Tapering on the Tolerability of DVS SR in Women With Vasomotor Symptoms Associated With Menopause: The PRIMMUS (PRIstiq for Managing Menopause and Understanding Symptoms) Study
Brief Title: The Effect Of Dose Titration And Dose Tapering On The Tolerability Of DVS SR In Women With Vasomotor Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3151A2-405
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Results first posted 2011-10-12 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Vasomotor Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- A (Active Comparator)
  Interventions: Drug: desvenlafaxine succinate sustained release
- B (Active Comparator)
  Interventions: Drug: desvenlafaxine succinate sustained release
- C (Active Comparator)
  Interventions: Drug: desvenlafaxine succinate sustained release
- D (Active Comparator)
  Interventions: Drug: desvenlafaxine succinate sustained release
- E (Active Comparator)
  Interventions: Drug: Placebo
- F (Active Comparator)
  Interventions: Drug: desvenlafaxine succinate sustained release
- G (Active Comparator)
  Interventions: Drug: desvenlafaxine succinate sustained release
- H (Placebo Comparator)
  Interventions: Drug: desvenlafaxine succinate sustained release

INTERVENTIONS:
Drug: desvenlafaxine succinate sustained release — Titration 100 mg
  Arms: A
Drug: desvenlafaxine succinate sustained release — Titration 50 mg
  Arms: B
Drug: desvenlafaxine succinate sustained release — Titration 25 mg, 50mg
  Arms: C
Drug: desvenlafaxine succinate sustained release — Titration 25 mg
  Arms: D
Drug: Placebo — Tapering placebo
  Arms: E
Drug: desvenlafaxine succinate sustained release — Tapering 50 mg, placebo
  Arms: F
Drug: desvenlafaxine succinate sustained release — Tapering 50 mg, 25 mg
  Arms: G
Drug: desvenlafaxine succinate sustained release — Tapering 50 mg QOD
  Arms: H

SUMMARY:
Desvenlafaxine succinate (DVS SR) is a serotonin and norepinephrine reuptake inhibitor (SNRI). It is a nonhormonal option for the treatment of Vasomotor Symptoms (VMS) associated with menopause. Nausea is the most common adverse event that is observed in clinical studies and is the main reason for discontinuation during the first week of therapy. Other adverse events (headache, nausea, and dizziness) associated with DVS SR have been noted to occur when subjects abruptly discontinue the medication. The purpose of this study is to evaluate several titration and tapering regimens of DVS SR to ensure a better tolerability profile at the start and completion of treatment. In addition, this study will provide a long posttreatment follow-up to assess any symptoms after treatment is discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, postmenopausal woman who seeks treatment for hot flushes.
* Meets 1 of the following: At least 12 months of spontaneous amenorrhea; At least 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) levels > 40 mIU/mL; At least 6 weeks postsurgical bilateral oophorectomy (with or without hysterectomy). Hysterectomized without bilateral oophorectomy and with serum FSH levels >40 mIU/mL.

Exclusion Criteria:

* History of a seizure disorder other than a single childhood febrile seizure.
* History or presence of clinically important hepatic or renal disease or other medical disease.
* Presence or recent history of major depressive disorder, bipolar disorder, psychotic disorder, or generalized anxiety disorder requiring therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2006-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (63):
- United States (47):
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Encinitas, California
  - Pfizer Investigational Site, Foothill Ranch, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Crystal River, Florida
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Idaho Falls, Idaho
  - Pfizer Investigational Site, Champaign, Illinois
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, South Bend, Indiana
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Canton, Michigan
  - Pfizer Investigational Site, Ypsilanti, Michigan
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Bismarck, North Dakota
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Watertown, South Dakota
  - Pfizer Investigational Site, Carrollton, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Hurst, Texas
  - Pfizer Investigational Site, Midland, Texas
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Seattle, Washington
- Canada (15):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Coquitlam, British Columbia
  - Pfizer Investigational Site, Langley, British Columbia
  - Pfizer Investigational Site, Surrey, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Newmarket, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Saint Romuald, Quebec
  - Pfizer Investigational Site, Shawinigan, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A2-405&StudyName=The%20Effect%20Of%20Dose%20Titration%20And%20Dose%20Tapering%20On%20The%20Tolerability%20Of%20DVS%20SR%20In%20Women%20With%20Vasomotor%20Symptoms

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 500 participants were randomized to the study, of which 7 were not treated due to other unspecified reasons. A second randomization occurred for the taper phase.
Groups:
- DVS 25 mg, Then 100 mg: Desvenlafaxine succinate (DVS) 25 milligram (mg) tablet taken orally daily for one week and placebo matched to 100 mg and 50 mg (double blind titration phase); then 100 mg for 15 week open label (OL) phase.
- DVS 25/50 mg, Then 100 mg: DVS 25 mg tablet taken orally for first 4 days followed by 50 mg for next 3 days for the first week and placebo matched to 100 mg (double blind titration phase); then 100 mg for 15 week OL phase.
- DVS 50 mg, Then 100 mg: DVS 50 mg tablet taken orally daily for one week and placebo matched to 100 mg and 25 mg (double blind titration phase); then 100 mg for 15 week OL phase.
- DVS 100 mg, Then 100 mg: DVS 100 mg tablet taken orally daily for one week and placebo matched to 25 mg and 50 mg (double blind titration phase); then 100 mg for 15 week OL phase.
- DVS 50 mg QOD: Re-randomized to DVS 50 mg tablet taken orally every other day (QOD) alternating with placebo matched to 50 mg QOD and placebo matched to 25 mg daily for 2 weeks (double blind tapering phase).
- DVS 50/25 mg: Re-randomized to DVS 50 mg tablet taken orally daily for first week along with placebo matched to 25 mg. For further 1 week, participants received DVS 25 mg tablet orally daily and placebo matched to 50 mg (double blind tapering phase).
- DVS 50 mg/Placebo: Re-randomized to DVS 50 mg tablet taken orally daily for first week and placebo matched to 25 mg. For further 1 week, participants received placebo matched to 25 mg and 50 mg (double blind tapering phase).
- Placebo: Re-randomized to placebo tablets matched to 25 mg and 50 mg taken orally daily for two weeks (double blind tapering phase).
Period: Double Blind Titration Phase
Arm/Group | DVS 25 mg, Then 100 mg | DVS 25/50 mg, Then 100 mg | DVS 50 mg, Then 100 mg | DVS 100 mg, Then 100 mg | DVS 50 mg QOD | DVS 50/25 mg | DVS 50 mg/Placebo | Placebo
Started | 126 | 121 | 124 | 122 | 0 | 0 | 0 | 0
Completed | 122 | 118 | 118 | 107 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 6 | 15 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 5 | 12 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Period: Between Titration and Open Label Phase
Arm/Group | DVS 25 mg, Then 100 mg | DVS 25/50 mg, Then 100 mg | DVS 50 mg, Then 100 mg | DVS 100 mg, Then 100 mg | DVS 50 mg QOD | DVS 50/25 mg | DVS 50 mg/Placebo | Placebo
Started | 122 | 118 | 118 | 107 | 0 | 0 | 0 | 0
Completed | 122 | 116 | 118 | 105 | 0 | 0 | 0 | 0
Not Completed | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Did not enter the open label phase | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Period: Open Label Phase
Arm/Group | DVS 25 mg, Then 100 mg | DVS 25/50 mg, Then 100 mg | DVS 50 mg, Then 100 mg | DVS 100 mg, Then 100 mg | DVS 50 mg QOD | DVS 50/25 mg | DVS 50 mg/Placebo | Placebo
Started | 122 | 116 | 118 | 105 | 0 | 0 | 0 | 0
Completed | 101 | 81 | 95 | 84 | 0 | 0 | 0 | 0
Not Completed | 21 | 35 | 23 | 21 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 14 | 6 | 7 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 7 | 5 | 4 | 0 | 0 | 0 | 0
Not completed — Other | 4 | 8 | 7 | 8 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Period: Double Blind Tapering Phase
Arm/Group | DVS 25 mg, Then 100 mg | DVS 25/50 mg, Then 100 mg | DVS 50 mg, Then 100 mg | DVS 100 mg, Then 100 mg | DVS 50 mg QOD | DVS 50/25 mg | DVS 50 mg/Placebo | Placebo
Started | 0 | 0 | 0 | 0 | 101 | 94 | 87 | 102
Completed | 0 | 0 | 0 | 0 | 97 | 90 | 80 | 95
Not Completed | 0 | 0 | 0 | 0 | 4 | 4 | 7 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4
Not completed — Investigator request | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DVS 25 mg, Then 100 mg: DVS 25 mg tablet taken orally daily for one week and placebo matched to 100 mg and 50 mg (double blind titration phase); then 100 mg for 15 week OL phase.
- Total: Total of all reporting groups
Arm/Group | DVS 25 mg, Then 100 mg | DVS 25/50 mg, Then 100 mg | DVS 50 mg, Then 100 mg | DVS 100 mg, Then 100 mg | Total
Number analyzed (Participants) | 126 | 121 | 124 | 122 | 493
Age Continuous [Mean (Standard Deviation); unit: Years] | 54.52 (5.01) | 54.40 (6.37) | 53.98 (5.16) | 53.48 (5.27) | 54.10 (5.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 121 | 124 | 122 | 493
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Nausea During the First 2 Weeks of Treatment
Description: Nausea by spontaneous reports to the investigators was counted if it was reported during first 2 weeks of treatment, and it was not seen before the first dose of treatment, or if it was seen before the first dose and the symptoms got worse. If multiple incidences occurred on the same participant during the 2 weeks, only 1 incidence was counted.
Time Frame: Baseline up to Week 2
Population: The titration population included all randomly assigned participants who had taken at least 1 dose of double-blind test article during the double-blind titration period.
Measure: Number; unit: Participants
Arm/Group | DVS 25 mg, Then 100 mg | DVS 25/50 mg, Then 100 mg | DVS 50 mg, Then 100 mg | DVS 100 mg, Then 100 mg
Number analyzed (Participants) | 126 | 121 | 124 | 122
Participants | 24 | 31 | 28 | 43
Statistical Analysis 1: Comparison: DVS 25 mg, Then 100 mg vs DVS 25/50 mg, Then 100 mg vs DVS 50 mg, Then 100 mg vs DVS 100 mg, Then 100 mg; Overall comparison was made between each titration regimen and the control regimen (100 mg); Test type: Superiority or Other; p = 0.024, Chi-squared — The analysis was done at a significance level of alpha = 0.05, 2-sided, without any adjustments for multiple comparisons

2. Primary Outcome: Discontinuation Emergent Signs and Symptoms (DESS) Total Score at the End of First Week of Tapering
Description: DESS: a clinician-administered 43-item assessment that evaluates discontinuation-emergent symptoms resulting from the withdrawal from test article. The DESS total score is the sum of the number of "new symptoms" and "old (but worse) symptoms" (1) and 0 for "old and unchanged symptom", "absent", or "old symptom but improved" for a total possible range of 0 to 43. A higher score indicates more symptoms.
Time Frame: Week 17
Population: The tapering population included all participants who had completed at least 6 weeks of treatment and taken at least 1 dose of double-blind test article during the tapering phase.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- DVS 50 mg QOD: Re-randomized to DVS 50 mg tablet taken orally QOD alternating with placebo matched to 50 mg QOD and placebo matched to 25 mg daily for 2 weeks (double blind tapering phase).
Arm/Group | DVS 50 mg QOD | DVS 50/25 mg | DVS 50 mg/Placebo | Placebo
Number analyzed (Participants) | 100 | 86 | 83 | 98
Units on a scale | 2.26 (3.46) | 2.28 (3.59) | 1.84 (3.36) | 7.07 (7.13)
Statistical Analysis 1: Comparison: DVS 50 mg QOD vs Placebo; For DVS 50 mg QOD, analysis of variance (ANOVA) was used to compare the DESS score between each tapering regimen and the control regimen (no tapering) for the titration population, where treatment was kept as the factor; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DVS 50/25 mg vs Placebo; For DVS 50/25 mg, ANOVA was used to compare the DESS score between each tapering regimen and the control regimen (no tapering) for the titration population, where treatment was kept as the factor; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: DVS 50 mg/Placebo vs Placebo; For DVS 50 mg/Placebo, ANOVA was used to compare the DESS score between each tapering regimen and the control regimen (no tapering) for the titration population, where treatment was kept as the factor; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: DESS Total Score at End of Second Week of Tapering
Description: as for outcome 2
Time Frame: Week 18
Population: Tapering population included all participants who had completed at least 6 weeks of treatment and taken at least 1 dose of double-blind test article during the tapering phase. Here, the 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure at the specified time point for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DVS 50 mg QOD | DVS 50/25 mg | DVS 50 mg/Placebo | Placebo
Number analyzed (Participants) | 89 | 87 | 79 | 91
Units on a scale | 1.19 (1.96) | 2.44 (5.53) | 4.46 (6.44) | 2.44 (4.96)
Statistical Analysis 1: Comparison: DVS 50 mg QOD vs Placebo; For DVS 50 mg QOD, ANOVA was used to compare the DESS score between each tapering regimen and the control regimen (no tapering) for the titration population, where treatment was kept as the factor; Test type: Superiority or Other; p = 0.092, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DVS 50/25 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.997, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: DVS 50 mg/Placebo vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.009, ANOVA — [p-value comment as in outcome 1, analysis 1]

4. Primary Outcome: DESS Total Score at 1 Week After the End of Tapering
Description: as for outcome 2
Time Frame: Week 19
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DVS 50 mg QOD | DVS 50/25 mg | DVS 50 mg/Placebo | Placebo
Number analyzed (Participants) | 59 | 57 | 47 | 59
Units on a scale | 3.22 (4.82) | 4.11 (5.77) | 1.70 (3.16) | 1.78 (3.20)
Statistical Analysis 1: Comparison: DVS 50 mg QOD vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.078, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DVS 50/25 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.005, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: DVS 50 mg/Placebo vs Placebo; For DVS 50mg/Placebo, ANOVA was used to compare the DESS score between each tapering regimen and the control regimen (no tapering) for the titration population, where treatment was kept as the factor; Test type: Superiority or Other; p = 0.929, ANOVA — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With Other Spontaneously Reported Adverse Events (AEs) in First 2 Weeks of Treatment
Description: Any untoward medical occurrence in a participant who received study drug was considered an AE, without regard to possibility of causal relationship.
Time Frame: Baseline up to Week 2
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | DVS 25 mg, Then 100 mg | DVS 25/50 mg, Then 100 mg | DVS 50 mg, Then 100 mg | DVS 100 mg, Then 100 mg
Number analyzed (Participants) | 126 | 121 | 124 | 122
Participants | 67 | 69 | 72 | 80

6. Secondary Outcome: Percentage of Participants Discontinuing Treatment Due to AEs in First 2 Weeks of Treatment
Description: as for outcome 5
Time Frame: Baseline up to Week 2
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | DVS 25 mg, Then 100 mg | DVS 25/50 mg, Then 100 mg | DVS 50 mg, Then 100 mg | DVS 100 mg, Then 100 mg
Number analyzed (Participants) | 126 | 121 | 124 | 122
Percentage of participants | 4.0 | 9.1 | 6.5 | 14.8
Statistical Analysis 1: Comparison: DVS 25 mg, Then 100 mg vs DVS 25/50 mg, Then 100 mg vs DVS 50 mg, Then 100 mg vs DVS 100 mg, Then 100 mg; Overall comparison was made between each titration regimen and the control regimen (100 mg); Test type: Superiority or Other; p = 0.017, Chi-squared — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants With Each DESS at the End of First Week of Tapering
Description: DESS: a clinician-administered 43-item assessment that evaluates discontinuation-emergent symptoms resulting from the withdrawal from test article.
Time Frame: Week 17
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | DVS 50 mg QOD | DVS 50/25 mg | DVS 50 mg/Placebo | Placebo
Number analyzed (Participants) | 101 | 94 | 87 | 102
Participants
  Agitation | 1 | 7 | 6 | 18
  Blurred vision | 4 | 4 | 2 | 13
  Bouts of crying or tearfulness | 5 | 3 | 6 | 24
  Burning, numbness, tingling sensations | 5 | 3 | 3 | 9
  Chills | 3 | 2 | 3 | 9
  Confusion or trouble concentrating | 5 | 4 | 2 | 21
  Diarrhea | 7 | 3 | 4 | 20
  Dizziness, lightheadedness, sensation of spinning | 18 | 7 | 9 | 41
  Elevated mood, feeling high | 1 | 0 | 0 | 13
  Fatigue, tiredness | 9 | 11 | 6 | 24
  Feeling unreal or detached | 6 | 2 | 1 | 20
  Fever | 2 | 0 | 1 | 4
  Forgetfulness or problems with memory | 6 | 6 | 3 | 12
  Headaches | 8 | 5 | 9 | 28
  Increased dreaming or nightmares | 14 | 13 | 12 | 35
  Increased saliva in mouth | 0 | 0 | 0 | 4
  Irritability | 6 | 6 | 6 | 26
  Mood swings | 4 | 5 | 4 | 19
  Muscle aches or pains | 5 | 8 | 3 | 19
  Muscle cramps, spasms, or twitching | 5 | 6 | 2 | 12
  Muscle tension or stiffness | 6 | 6 | 7 | 18
  Nausea | 14 | 7 | 5 | 28
  Nervousness or anxiety | 2 | 5 | 7 | 19
  Nose running | 3 | 3 | 3 | 7
  Problems with speech or speaking clearly | 3 | 2 | 0 | 6
  Restless feeling in legs | 5 | 4 | 0 | 4
  Ringing or noises in the ears | 6 | 2 | 6 | 14
  Shaking, trembling | 4 | 4 | 2 | 11
  Shortness of breath, gasping for air | 1 | 3 | 1 | 6
  Sore eyes | 3 | 3 | 5 | 8
  Stomach bloating | 5 | 6 | 5 | 19
  Stomach cramps | 6 | 4 | 0 | 11
  Sudden outbursts of anger | 3 | 4 | 2 | 11
  Sudden panic or anxiety attacks | 0 | 2 | 0 | 9
  Sudden worsening of mood | 3 | 6 | 4 | 22
  Sweating more than usual | 23 | 19 | 14 | 44
  Trouble sleeping, insomnia | 13 | 11 | 8 | 37
  Uncontrolled mouth/tongue movements | 1 | 1 | 0 | 0
  Unsteady gait or incoordination | 4 | 1 | 0 | 16
  Unusual sensitivity to sound | 1 | 5 | 1 | 7
  Unusual tastes or smells | 1 | 2 | 1 | 4
  Unusual visual sensations | 1 | 0 | 0 | 10
  Vomiting | 4 | 1 | 0 | 11

8. Secondary Outcome: Number of Participants With Each DESS at the End of Second Week of Tapering
Description: as for outcome 7
Time Frame: Week 18
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | DVS 50 mg QOD | DVS 50/25 mg | DVS 50 mg/Placebo | Placebo
Number analyzed (Participants) | 89 | 87 | 79 | 91
Participants
  Agitation | 6 | 4 | 10 | 9
  Blurred vision | 2 | 6 | 7 | 3
  Bouts of crying or tearfulness | 2 | 5 | 18 | 6
  Burning, numbness, tingling sensations | 0 | 2 | 3 | 4
  Chills | 1 | 3 | 8 | 4
  Confusion or trouble concentrating | 0 | 7 | 11 | 4
  Diarrhea | 2 | 2 | 5 | 1
  Dizziness, lightheadedness, sensation of spinning | 2 | 12 | 21 | 7
  Elevated mood, feeling high | 3 | 3 | 5 | 3
  Fatigue, tiredness | 3 | 12 | 14 | 11
  Feeling unreal or detached | 0 | 5 | 9 | 3
  Fever | 0 | 0 | 1 | 1
  Forgetfulness or problems with memory | 1 | 6 | 4 | 2
  Headaches | 4 | 5 | 8 | 4
  Increased dreaming or nightmares | 4 | 5 | 10 | 8
  Increased saliva in mouth | 1 | 1 | 2 | 4
  Irritability | 5 | 10 | 18 | 13
  Mood swings | 3 | 7 | 14 | 5
  Muscle aches or pains | 2 | 8 | 9 | 7
  Muscle cramps, spasms, or twitching | 7 | 3 | 6 | 5
  Muscle tension or stiffness | 1 | 8 | 7 | 7
  Nausea | 3 | 6 | 15 | 4
  Nervousness or anxiety | 4 | 6 | 12 | 8
  Nose running | 1 | 5 | 4 | 7
  Problems with speech or speaking clearly | 0 | 3 | 4 | 1
  Restless feeling in legs | 4 | 4 | 4 | 4
  Ringing or noises in the ears | 1 | 4 | 6 | 2
  Shaking, trembling | 1 | 3 | 3 | 3
  Shortness of breath, gasping for air | 0 | 2 | 1 | 4
  Sore eyes | 2 | 4 | 3 | 5
  Stomach bloating | 1 | 5 | 6 | 5
  Stomach cramps | 2 | 3 | 4 | 0
  Sudden outbursts of anger | 4 | 5 | 12 | 8
  Sudden panic or anxiety attacks | 0 | 3 | 5 | 1
  Sudden worsening of mood | 6 | 5 | 18 | 8
  Sweating more than usual | 19 | 17 | 23 | 23
  Trouble sleeping, insomnia | 8 | 9 | 22 | 19
  Uncontrolled mouth/tongue movements | 0 | 1 | 0 | 1
  Unsteady gait or incoordination | 0 | 7 | 5 | 3
  Unusual sensitivity to sound | 0 | 5 | 3 | 2
  Unusual tastes or smells | 1 | 1 | 4 | 1
  Unusual visual sensations | 0 | 0 | 3 | 2
  Vomiting | 0 | 0 | 5 | 0

9. Secondary Outcome: Number of Participants With Each DESS One Week After End of Tapering
Description: as for outcome 7
Time Frame: Week 19
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | DVS 50 mg QOD | DVS 50/25 mg | DVS 50 mg/Placebo | Placebo
Number analyzed (Participants) | 59 | 57 | 47 | 59
Participants
  Agitation | 6 | 4 | 6 | 5
  Blurred vision | 2 | 0 | 0 | 1
  Bouts of crying or tearfulness | 7 | 7 | 2 | 3
  Burning, numbness, tingling sensations | 2 | 9 | 0 | 2
  Chills | 3 | 3 | 1 | 3
  Confusion or trouble concentrating | 6 | 7 | 4 | 2
  Diarrhea | 3 | 3 | 1 | 1
  Dizziness, lightheadedness, sensation of spinning | 13 | 17 | 2 | 0
  Elevated mood, feeling high | 1 | 2 | 0 | 0
  Fatigue, tiredness | 9 | 10 | 2 | 8
  Feeling unreal or detached | 6 | 5 | 1 | 3
  Fever | 2 | 0 | 0 | 0
  Forgetfulness or problems with memory | 5 | 3 | 2 | 3
  Headaches | 4 | 11 | 3 | 5
  Increased dreaming or nightmares | 7 | 10 | 0 | 3
  Increased saliva in mouth | 0 | 1 | 1 | 1
  Irritability | 11 | 9 | 7 | 6
  Mood swings | 4 | 5 | 6 | 4
  Muscle aches or pains | 5 | 8 | 5 | 3
  Muscle cramps, spasms, or twitching | 5 | 5 | 1 | 1
  Muscle tension or stiffness | 5 | 9 | 3 | 2
  Nausea | 5 | 5 | 0 | 1
  Nervousness or anxiety | 9 | 10 | 5 | 3
  Nose running | 1 | 2 | 3 | 1
  Problems with speech or speaking clearly | 0 | 2 | 0 | 0
  Restless feeling in legs | 1 | 6 | 3 | 1
  Ringing or noises in the ears | 3 | 8 | 0 | 0
  Shaking, trembling | 3 | 3 | 0 | 1
  Shortness of breath, gasping for air | 1 | 1 | 1 | 0
  Sore eyes | 3 | 4 | 1 | 2
  Stomach bloating | 3 | 4 | 1 | 4
  Stomach cramps | 2 | 3 | 0 | 2
  Sudden outbursts of anger | 4 | 3 | 3 | 5
  Sudden panic or anxiety attacks | 1 | 5 | 2 | 2
  Sudden worsening of mood | 7 | 4 | 5 | 5
  Sweating more than usual | 21 | 19 | 4 | 12
  Trouble sleeping, insomnia | 12 | 13 | 5 | 7
  Uncontrolled mouth/tongue movements | 0 | 1 | 0 | 0
  Unsteady gait or incoordination | 4 | 5 | 0 | 1
  Unusual sensitivity to sound | 1 | 2 | 0 | 1
  Unusual tastes or smells | 1 | 3 | 0 | 0
  Unusual visual sensations | 0 | 3 | 0 | 1
  Vomiting | 1 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Showing Satisfaction With Tolerability During the First Two Weeks of Treatment
Description: Satisfaction with tolerability (lack of bothersomeness) was assessed using a questionnaire via an interactive voice response system (IVRS)/interactive web based response system (IWRS), and evaluated based on participants' response of extremely satisfied, satisfied, neutral, dissatisfied or extremely dissatisfied with the study medication.
Time Frame: Week 1 and Week 2
Population: The titration population included all randomly assigned participants who had taken at least 1 dose of double-blind test article during the double-blind titration period. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the time points for each group respectively.
Measure: Number; unit: Participants
Arm/Group | DVS 25 mg, Then 100 mg | DVS 25/50 mg, Then 100 mg | DVS 50 mg, Then 100 mg | DVS 100 mg, Then 100 mg
Number analyzed (Participants) | 126 | 121 | 124 | 122
Participants
  Week 1: Extremely dissatisfied (n=124,119,120,111) | 2 | 3 | 1 | 4
  Week 1: Dissatisfied (n=124,119,120,111) | 1 | 6 | 8 | 16
  Week 1: Neutral (n=124,119,120,111) | 20 | 13 | 28 | 19
  Week 1: Satisfied (n=124,119,120,111) | 47 | 48 | 43 | 39
  Week 1: Extremely satisfied (n=124,119,120,111) | 54 | 49 | 40 | 33
  Week 2: Extremely dissatisfied (n=115,105,113,94) | 2 | 0 | 0 | 0
  Week 2: Dissatisfied (n=115,105,113,94) | 3 | 4 | 8 | 1
  Week 2: Neutral (n=115,105,113,94) | 17 | 17 | 18 | 15
  Week 2: Satisfied (n=115,105,113,94) | 43 | 35 | 41 | 40
  Week 2: Extremely satisfied (n=115,105,113,94) | 50 | 49 | 46 | 38

11. Secondary Outcome: Number of Participants Showing Satisfaction With Tolerability at the End of Tapering
Description: Satisfaction with tolerability (lack of bothersomeness) was assessed using a questionnaire via an IVRS/IWRS and evaluated based on participants' response of extremely satisfied, satisfied, neutral, dissatisfied or extremely dissatisfied with the study medication.
Time Frame: Week 19
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | DVS 50 mg QOD | DVS 50/25 mg | DVS 50 mg/Placebo | Placebo
Number analyzed (Participants) | 53 | 52 | 40 | 55
Participants
  Extremely dissatisfied | 7 | 5 | 3 | 6
  Dissatisfied | 10 | 7 | 3 | 5
  Neutral | 10 | 5 | 5 | 7
  Satisfied | 16 | 23 | 19 | 19
  Extremely satisfied | 10 | 12 | 10 | 18

12. Secondary Outcome: Menopause Symptoms-treatment Satisfaction Questionnaire (MS-TSQ) Score
Description: MS-TSQ is a questionnaire assessing participants' degree of satisfaction with regard to the test article which was administered to the participants via an IVRS/IWRS. The questionnaire comprised 8 questions and each was rated on a scale from 0 (extremely dissatisfied) to 4 (extremely satisfied).
Time Frame: Week 16
Population: The OL population included all participants who had taken at least 1 dose of open label test article. Here, the 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure at the specified time point for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- DVS 100 mg: DVS 100 mg tablet taken orally daily for 15 weeks (OL phase).
Arm/Group | DVS 100 mg
Number analyzed (Participants) | 270
Units on a scale
  Ability to control hot flushes during the day | 2.64 (1.19)
  Ability to control hot flushes during the night | 2.71 (1.26)
  Effect on quality of sleep | 2.59 (1.18)
  Effect on mood or emotions | 3.02 (0.86)
  Effect on interest in sex | 2.37 (1.00)
  Effect on ability to concentrate | 2.67 (0.84)
  Tolerability to side effects | 3.04 (0.94)
  Overall satisfaction | 2.81 (1.10)

13. Secondary Outcome: Change From Baseline in Menopause-specific Quality of Life Questionnaire (MenQOL) Score at Week 4, Week 8, Week 12 and Week 16
Description: MenQOL questionnaire assessed how bothered participants were with 31 symptoms. It contains domains: vasomotor (items 1-3); psychosocial (items 4-10); physical (items 11-26); sexual (items 27-29); in addition to nausea and indigestion. 31 individual symptoms are rated on a scale of 0 (not at all bothered) to 6 (extremely bothered). Total possible score ranged from 0 to 186. MenQOL summary score was calculated as mean of four domain scores (Physical function, Psychosocial function, Sexual function and Vasomotor function) ranging from 1 to 8, with higher scores indicating worse quality of life.
Time Frame: Baseline, Week 4, Week 8, Week 12 and Week 16
Population: The OL population included all participants who had taken at least 1 dose of open label test article. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the time points for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DVS 100 mg
Number analyzed (Participants) | 406
Units on a scale
  Baseline | 4.46 (1.20)
  Week 4 (n=385) | 2.99 (1.09)
  Week 8 (n=364) | 2.85 (1.08)
  Week 12 (n=354) | 2.76 (1.06)
  Week 16 (n=277) | 2.67 (1.17)
Statistical Analysis 1: Comparison: DVS 100 mg; Comparison was made between the difference in the means from the baseline value and post-baseline (Week 4) value with 0; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DVS 100 mg; Comparison was made between the difference in the means from the baseline value and post-baseline (Week 8) value with 0; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: DVS 100 mg; Comparison was made between the difference in the means from the base value and post-baseline (Week 12) value with 0; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: DVS 100 mg; Comparison was made between the difference in the means from the baseline value and post-baseline (Week 16) value with 0; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

14. Other Pre Specified Outcome: Mean Age of the Participants in Tapering Phase
Description: Participants were re-randomized to tapering phase after OL phase.
Time Frame: Week 17
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | DVS 50 mg QOD | DVS 50/25 mg | DVS 50 mg/Placebo | Placebo
Number analyzed (Participants) | 101 | 94 | 87 | 102
Years | 53.72 (5.02) | 54.56 (5.21) | 54.20 (6.31) | 54.14 (5.09)

15. Other Pre Specified Outcome: Gender of the Participants in Tapering Phase
Description: Participants were re-randomized to tapering phase after OL phase.
Time Frame: Week 17
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | DVS 50 mg QOD | DVS 50/25 mg | DVS 50 mg/Placebo | Placebo
Number analyzed (Participants) | 101 | 94 | 87 | 102
Participants
  Female | 101 | 94 | 87 | 102
  Male | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- DVS 25 mg (Titration Phase): DVS 25 mg tablet taken orally daily for one week and placebo matched to 100 mg and 50 mg (double blind titration phase).
- DVS 25/50 mg (Titration Phase): DVS 25 mg tablet taken orally for first 4 days followed by 50 mg for next 3 days for the first week and placebo matched to 100 mg (double blind titration phase).
- DVS 50 mg (Titration Phase): DVS 50 mg tablet taken orally daily for one week and placebo matched to 100 mg and 25 mg (double blind titration phase).
- DVS 100 mg (Titration Phase): DVS 100 mg tablet taken orally daily for one week and placebo matched to 25 mg and 50 mg (double blind titration phase).
- DVS 100 mg (OL Phase): After 1 week of double blind titration phase, DVS 100 mg tablet taken orally daily for 15 weeks.
- DVS 50 mg QOD (Tapering Phase): Re-randomized to DVS 50 mg tablet taken orally QOD alternating with placebo matched to 50 mg QOD and placebo matched to 25 mg daily for 2 weeks (double blind tapering phase).
- DVS 50/25 mg (Tapering Phase): Re-randomized to DVS 50 mg tablet taken orally daily for first week along with placebo matched to 25 mg. For further 1 week, participants received DVS 25 mg tablet orally daily and placebo matched to 50 mg (double blind tapering phase).
- DVS 50 mg/Placebo (Tapering Phase): Re-randomized to DVS 50 mg tablet taken orally daily for first week and placebo matched to 25 mg. For further 1 week, participants received placebo matched to 25 mg and 50 mg (double blind tapering phase).
- Placebo (Tapering Phase): Re-randomized to placebo tablets matched to 25 mg and 50 mg taken orally daily for two weeks (double blind tapering phase).
Arm/Group | DVS 25 mg (Titration Phase) | DVS 25/50 mg (Titration Phase) | DVS 50 mg (Titration Phase) | DVS 100 mg (Titration Phase) | DVS 100 mg (OL Phase) | DVS 50 mg QOD (Tapering Phase) | DVS 50/25 mg (Tapering Phase) | DVS 50 mg/Placebo (Tapering Phase) | Placebo (Tapering Phase)
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/121 | 0/124 | 0/122 | 3/461 | 0/101 | 0/94 | 0/87 | 1/102
Other Adverse Events (participants affected / at risk) | 50/126 | 55/121 | 57/124 | 73/122 | 340/461 | 74/101 | 64/94 | 67/87 | 79/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DVS 25 mg (Titration Phase) (N=126) | DVS 25/50 mg (Titration Phase) (N=121) | DVS 50 mg (Titration Phase) (N=124) | DVS 100 mg (Titration Phase) (N=122) | DVS 100 mg (OL Phase) (N=461) | DVS 50 mg QOD (Tapering Phase) (N=101) | DVS 50/25 mg (Tapering Phase) (N=94) | DVS 50 mg/Placebo (Tapering Phase) (N=87) | Placebo (Tapering Phase) (N=102)
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DVS 25 mg (Titration Phase) (N=126) | DVS 25/50 mg (Titration Phase) (N=121) | DVS 50 mg (Titration Phase) (N=124) | DVS 100 mg (Titration Phase) (N=122) | DVS 100 mg (OL Phase) (N=461) | DVS 50 mg QOD (Tapering Phase) (N=101) | DVS 50/25 mg (Tapering Phase) (N=94) | DVS 50 mg/Placebo (Tapering Phase) (N=87) | Placebo (Tapering Phase) (N=102)
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 1 | 2 | 20 | 6 | 3 | 1 | 5
Accidental injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 18 | 2 | 2 | 3 | 5
Asthenia (General disorders) | 6 | 4 | 12/121 | 11 | 55 | 14 | 5 | 5 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 24 | 1 | 3 | 4 | 2
Chills (General disorders) | 1 | 0 | 2 | 5 | 0 | 0 | 3 | 2 | 4 (102)
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Flu syndrome (General disorders) | 0 | 0 | 0 | 0 | 13 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 15 | 12 | 14 | 14 | 77 | 12 | 9 | 11 | 19
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 23 | 2 | 3 | 3 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 10 | 2 | 3 | 3 | 2
Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 20 | 4 | 5 | 1 | 4
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 7
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Palpitation (Cardiac disorders) | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 4
Vasodilatation (Vascular disorders) | 0 | 0 | 0 | 0 | 16 | 7 | 6 | 2 | 12
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 26 | 7 | 8 | 5 | 6
Anorexia (Gastrointestinal disorders) | 1 | 2 | 5 | 4 | 16 | 1 | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 5 | 4 | 7 | 42 | 6 | 5 | 4 | 5
Diarrhea (Gastrointestinal disorders) | 3 | 4 | 1 | 1 | 24 | 6 | 4 | 5 | 10
Dry mouth (Gastrointestinal disorders) | 4 | 9 | 11 | 18 | 44 | 6 | 4 | 3 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 3 | 5 | 19 | 3 | 3 | 2 | 3
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Increased appetite (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Increased salivation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 19 | 26 | 26 | 41 | 91 | 14 | 13 | 8 | 12
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3 | 4 | 0 | 5 | 1 | 2 | 4
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Echymosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Hypercholesteremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 3
Hyperlipemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 21 | 1 | 4 | 5 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 19 | 4 | 3 | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 24 | 7 | 5 | 1 | 7
Abnormal dreams (Nervous system disorders) | 0 | 0 | 0 | 0 | 45 | 11 | 15 | 10 | 15
Agitation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 4
Anxiety (Nervous system disorders) | 2 | 4 | 1 | 0 | 17 | 1 | 5 | 3 | 7
Confusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
Depersonalization (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 5
Dizziness (Nervous system disorders) | 2 | 6 | 5 | 11 | 45 | 16 | 16 | 13 | 16
Emotional lability (Nervous system disorders) | 0 | 0 | 0 | 0 | 12 | 4 | 2 | 5 | 10
Euphoria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Hostility (Nervous system disorders) | 0 | 0 | 0 | 0 | 13 | 2 | 2 | 3 | 4
Hypesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 10 | 0 | 2 | 2 | 3
Incoordination (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 6
Insonmnia (Nervous system disorders) | 3 | 7 | 7 | 6 | 62 | 14 | 10 | 8 | 13
Libido decreased (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Memory impairement (Nervous system disorders) | 0 | 0 | 0 | 0 | 17 | 6 | 0 | 4 | 3
Nervousness (Nervous system disorders) | 2 | 3 | 0 | 2 | 12 | 1 | 2 | 3 | 3
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 19 | 2 | 4 | 4 | 4
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 19 | 5 | 8 | 2 | 5
Somnolence (Nervous system disorders) | 0 | 2 | 7 | 15 | 31 | 2 | 2 | 3 | 4
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1
Thinking abnormal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 2 | 3 | 3 | 14 | 3 | 3 | 1 | 3
Vertigo (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 2 | 3 | 2 | 3
Cough increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 3
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 19 | 0 | 0 | 0 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 22 | 3 | 9 | 4 | 3
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 14 | 2 | 1 | 0 | 3
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 12 | 0 | 1 | 2 | 1
Sweating (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 43 | 8 | 11 | 10 | 18
Abnormal vision (Eye disorders) | 1 | 1 | 2 | 4 | 20 | 3 | 6 | 5 | 6
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 3
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Taste perversion (Nervous system disorders) | 0 | 0 | 0 | 0 | 16 | 2 | 4 | 2 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 13 | 3 | 4 | 3 | 6
Abnormal ejaculation /orgasm (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Reaction unevaluable (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.